CLINICAL TRIAL: NCT03712267
Title: Electronic Media and Its Application in Psychotherapy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mclean Hospital (Other)
Collaborators: Once Upon a Time Foundation (Other)
Responsible Party: Principal Investigator, Ipsit Vihang Vahia, Medical Director, Geriatric Psychiatry Outpatient Programs, Mclean Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 2018P002179
Record Dates: First submitted 2018-10-12; First posted 2018-10-19 (Actual); Last update posted 2025-11-05 (Actual); Status verified 2025-11

CONDITIONS: Anxiety Disorders; Depression; Electronic Media
MeSH Terms: conditions — Anxiety Disorders; Depression | interventions — Therapeutics

STUDY DESIGN:
Who Masked: Participant
Masking Description: Study participants will be randomized to either the intervention group or the control group through an online computer randomizing generator. This is not a blinded randomized control trial.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Electronic Media Enhanced (Experimental): Research assistants will collect information on participants' electronic messaging behavior and content and provide that for use to participants' clinicians.
  Interventions: Behavioral: Electronic Media Enhanced
- Treatment As Usual (Placebo Comparator): Participants will not have their electronic messaging reviewed prior to their typically scheduled clinical appointments.
  Interventions: Behavioral: Treatment as Usual

INTERVENTIONS:
Behavioral: Electronic Media Enhanced — Research assistants will provide participants' therapists with information from participants' electronic messaging prior to typically scheduled clinical appointments.
  Arms: Electronic Media Enhanced
Behavioral: Treatment as Usual — Research assistants will not review or provide participants' therapists with information from participants' electronic media and will compare with the Electronic Media Enhanced cohort to see if there was a difference in therapy outcomes.
  Arms: Treatment As Usual

SUMMARY:
This randomized control trial aims to establish whether viewing and discussing patients' electronic communication (texts, emails, Facebook direct messaging, etc) impacts clinical care and decision making across the lifespan.

DETAILED DESCRIPTION:
This study explores the usefulness and effectiveness of including electronic communication as part of standard clinical care. Participants will provide information and content from their electronic media to research assistants during in person interviews if they are in the intervention group. Research assistants will then give clinicians the information collected, so the clinicians can incorporate the data into the session as they see fit. Therapists will retain full clinical discretion of how they continue to conduct their therapy sessions. The investigators will compare the impact of receiving this electronic enhancement intervention versus only receiving treatment as usual care on mental health related functioning and therapeutic alliance.

ELIGIBILITY:
Inclusion Criteria:

1. Are currently receiving psychotherapy at McLean and have had at least 4 visits with their current therapy provider in outpatient clinics or 2 sessions with their therapy provider in partial hospitalization or residential settings
2. Age 18-85, and fluent in English
3. Have a primary diagnosis of anxiety or depression (as determined by self-report and review of medical records, which should list a primary depression or anxiety spectrum diagnosis). Symptomatology can be active or in remission.
4. Are actively using at least 1 platform for text messaging (i.e. they should have an account on each platform and have produced content within the month prior to beginning the study). This will be based on self report.
5. Use a mobile device for text messaging
6. Able to provide informed consent.

Exclusion Criteria:

1. Probable or diagnosed dementia or cognitive impairment, or neurodevelopmental disorder (such as an autism spectrum disorder) based on self report and review of medical records.

   - Individuals with Attention-Deficit/Hyperactivity Disorder (ADHD) or Attention-Deficit Disorder (ADD) may be eligible provided symptoms have been stable for at least 6 months.
2. Active psychotic symptoms

   - History of psychosis is allowable only if the patient has not had symptoms for at least a year
3. Are actively receiving ECT treatment
4. Current alcohol or drug abuse problem (based on self report and review of medical records)

   - History of substance use is fine, provided there has been no relapse or withdrawal symptoms in the month leading up to enrollment
5. Are involuntarily admitted to McLean Hospital

Ages: 14 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 110 (Actual)
Dates: Start 2018-12-13 (Actual); Primary Completion 2023-08-31 (Actual); Study Completion 2023-08-31 (Actual)

PRIMARY OUTCOMES:
Improvement in Mental Health Related Quality of Life/Functioning | After final visit
  Investigators will use the Short Form Health - 36 Item Survey (SF-36) to assess whether use of electronic media will lead to participants reporting improved functioning/quality of life. The SF-36 is a patient-administered scale and focuses on 8 domains including social functioning, perceptions of health, emotional well-being, role limitations due to physical or emotional concerns, and physical functioning.
Therapeutic Alliance | After final visit
  Investigators will use the Working Alliance Inventory - Short Revised (WAI-SR) scale to assess whether use of electronic media will lead to participants reporting an enhanced working alliance. The working alliance inventory is a 12 item measure of the client's/patient's perception of how comfortable they believe their alliance with their therapist is. Each item is rated on a scale of 1-5, and measures how frequently participants believe criteria has been achieved. A score of 1 typically represents that the specific item has been achieved least frequently and a sore of 5 indicates that the specific item is achieved at every session. The items are then summed up to compute a total score.

SECONDARY OUTCOMES:
Clinical Outcome - Improvement in scores of depression | Every 4 visits, up to 13 visits
  Investigators will use the Patient Health Questionnaire-9 (OHQ-9) to assess changes in patient's/client's symptoms of depression. The Patient Health Questionnaire-9 is a 9 item questionnaire used to screen for symptoms of major depression. It is self-administered by participants. Items are scored on a scale of 0-3 with total scores ranging from 0-27. Higher scores indicate more severe depressive symptoms.
Clinical Outcome - Improvement in scores of anxiety | Every 4 visits, up to 13 visits
  Investigators will use the General Anxiety Disorder Scale (GAD-7) to assess changes in patient's/client's symptoms of anxiety. The Generalized Anxiety Disorder Scale is a 7-item questionnaire used to screen symptoms of anxiety disorders. It is self-administered by the participant. The 7 items are scored on a 0-3 scale, and total scores range from 0-21. Higher scores indicate more severe anxiety symptoms.

CONTACTS AND LOCATIONS:
Overall Officials: Ipsit Vahia, MD, Principal Investigator — Mclean Hospital; Kerry Ressler, MD; PhD, Principal Investigator — Mclean Hospital
Locations (1):
- McLean Hospital, Belmont, Massachusetts, United States